CLINICAL TRIAL: NCT03134690
Title: Evaluation of a Novel " Delayed Start" Protocol With Gonadotropin-releasing Hormone Antagonist in Poor Responders: A Randomized Clinical Trial Phase 3
Brief Title: GnRh Antagonist Protocol With Delayed Start Stimulation in Patients With Poor Ovarian Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Emb-028
Record Dates: First submitted 2016-12-19; First posted 2017-05-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Infertility, Female
Keywords: Poor ovarian response gonadotropins antagonist
MeSH Terms: conditions — Infertility, Female | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- delayed start antagonist (Experimental): 60 women with poor ovarian responses undergo ovarian stimulation with delayed start antagonist.
  Interventions: Procedure: delayed start
- conventional antagonist (Experimental): 60 women with diagnose of poor ovarian response will have undergone ovarian stimulation with conventional antagonist protocol.
  Interventions: Procedure: Conventional

INTERVENTIONS:
Procedure: delayed start — In this protocol, ovarian stimulation will be started from ninth day of menstrual cycle .
  Arms: delayed start antagonist
Procedure: Conventional — In this protocol, ovarian stimulation will be started from the 2th or 3th day of the menstrual cycle.
  Arms: conventional antagonist

SUMMARY:
The main outcome measures are the number of dominant follicles (≥13 mm) on the day of hCG trigger and the number of mature (MII) oocytes collected after conventional versus delayed-start ovarian stimulation protocol. Secondary outcome measures are including total number of oocytes retrieved, oocyte maturity rate (number of MII oocytes/total number of oocytes), oocyte yield (total number of oocytes retrieved/ antral follicle count [AFC]), mature oocyte yield (number of mature oocytes retrieved/AFC), total dosage of gonadotropin (recombinant FSH and/or highly purified hMG) needed, number of days needed for ovarian stimulation, quality of obtained embryos, fertilization rate (the proportion of total number of two-pronuclear [2PN] stage zygotes /per total injected MII oocytes), implantation rate (total number of observed gestational sac/ number of transferred embryos) and clinical pregnancy rate (presence of fetal heart beat by transvaginal ultrasound per embryo transfer).

DETAILED DESCRIPTION:
One of the principal steps to obtain the favorable success is still related to the number of retrieved oocytes after hormonal stimulation by gonadotropins in combination with GnRH analogues. In the patients with "poor ovarian response" diagnosis, the limited number of obtained oocytes remains the main obstacle in optimizing the live birth rates. The objective of present study is to evaluate a new procedure to increase a cohort of the growing antral follicles and consequently the number of retrieved oocytes after hormonal stimulation by gonadotropins in combination with GnRH antagonist. In present study, eligible patients with diagnosis poor ovarian responder based on the Bologna criteria are included. Ovarian stimulation procedure will be performed by antagonist protocol. All the patients will be received two tablets daily of Estradiol valerate (Estraval®, 2 mg, Aburaihan Co., Tehran, Iran) starting a week after LH surge until menses. The hormonal evaluation (serum LH and FSH) and basic vaginal ultrasound will be performed before the starting ovarian stimulation on the 2th or 3th day of the menstrual cycle. On this day, the block randomization method will be designed to randomize allocation of patients into groups with blocks of size 4.

In the Group A: treatment with GnRH antagonists (Cetrotide®, 0.25 mg cetrorelix acetate, Serono, Inc) will be started on the 2th or 3th day of the menstrual cycle and continues until the ninth day. Then, the ovarian stimulation with gonadotropin 300 IU recombinant FSH (Gonal - F®, Serono Laboratories Ltd, Geneva, Switzerland) and 150 IU of hMG (Menopur®; Ferring) will be started from ninth day of menstrual cycle until the day of hCG administration. The monitoring of ovarian stimulation will be done every other day by vaginal ultrasound and whenever at least 1 to 3 follicles larger than 13 mm are observed, the antagonist injection (Cetrotide®, 0.25 mg cetrorelix acetate, Serono, Inc) will be started again to prevent premature LH surge and continues until the prescription of hCG. When at least two follicles greater than 17 to 18 mm is seen, two pre-filled syringes of recombinant human chorionic gonadotropin (rhCG) (Ovitrelle®, 250 μg/0.5 ml, Merck, Serono, Inc) will be administered. The patients will undergo puncture operation 32-34 hours after hCG injection.

In the control group (B), as conventional antagonist procedure, the ovarian stimulation with gonadotropin 300 IU recombinant FSH (Gonal - F®, Serono Laboratories Ltd, Geneva, Switzerland) and 150 IU of hMG ( Menopur®; Ferring ) will be started from on the 2th or 3th day of the menstrual cycle. The monitoring of ovarian stimulation will be done every other day by vaginal ultrasound and whenever at least 1 to 3 follicles larger than 13 mm are observed, the antagonist injection (Cetrotide®, 0.25 mg cetrorelix acetate, Serono, Inc) will be started again to prevent premature LH surge and continues until the prescription of rhCG. 32-34 hours after the rhCG injection, the ovum pick up will be performed and subsequently intracytoplasmic sperm injection (ICSI) /in-vitro fertilization (IVF) will be done for all the patients.

ELIGIBILITY:
Poor ovarian response is defined according to the Bologna criteria and existence of at least two of the following criteria:

1. a previous history of POR (retrieved oocytes ≤3) in a conventional stimulation protocol,
2. advanced maternal age (≥40 years) or any other risk factors for POR (e.g. a history of ovarian surgery)
3. abnormal ovarian reserve test (i.e. antral follicle count (AFC) < 5 follicles or anti-Mȕllerian hormone (AMH) < 1.1 ng/ml)

Exclusion Criteria:

1. Premature ovarian failure (basal follicle stimulating hormone (FSH) above 20 IU/l or no antral follicle in ultrasound examination),
2. ِDonor/recipient treatments,
3. Metabolic or endocrine disorders including hyperprolactinoma and hypo/hyperthyroidism, endometriosis,
4. Body mass index > 30 kg/m2,
5. azoospermic male partner.
6. A minimum of 2 or more month's interval from the previous ovarian stimulation is considered to prevent any potential source of error.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-01; Primary Completion 2018-04 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
number of dominant follicles (≥13 mm) | 24h after rhCG injection
  The number of dominant follicles (≥13 mm) on the day of hCG trigger
Total number of oocytes | 32-34 hours after rhCG
  the number of mature oocytes collected after conventional versus delayed-start ovarian stimulation protocol

SECONDARY OUTCOMES:
Total number of retrieved oocytes | 32-34 hours after rhCG injection
  Total number of retrieved oocytes 32-34 hours after rhCG injection .
Quality of obtained embryos | on the third day after oocyte retrieval
  we score embryo quality according to the following quality criteria: Excellent (Day 3: 6-8 even size blastomeres with ≤10% fragmentation), Good (Day 3: 6-8 even or uneven size blastomeres with 10%-20% fragmentation), Poor (Uneven and few blastomeres with >20% fragmentation)

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Mahnaz Ashrafi, MD, Study Director — Department of Endocrinology and Female Infertility, Reproductive Biomedicine Research Center, ACECR, Tehran, Iran; Mandana Hemmat, MD, Principal Investigator — Department of Endocrinology and Female Infertility, Reproductive Biomedicine Research Center, ACECR, Tehran, Iran; Arezoo Arabipour, MSc, Principal Investigator — Department of Endocrinology and Female Infertility, Reproductive Biomedicine Research Center, ACECR, Tehran, Iran
Locations (1):
- Royan Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ashrafi M, Arabipoor A, Yahyaei A, Zolfaghari Z, Ghaffari F. Does the "delayed start" protocol with gonadotropin-releasing hormone antagonist improve the pregnancy outcome in Bologna poor responders? a randomized clinical trial. Reprod Biol Endocrinol. 2018 Dec 28;16(1):124. doi: 10.1186/s12958-018-0442-y. PMID 30593268